CLINICAL TRIAL: NCT01531387
Title: Sparing Conversion to Abnormal TCD Elevation (SCATE) - a Phase III Clinical Trial to Compare Standard Care (Observation) With Alternative Therapy (Hydroxyurea) for Reducing the Risk of Converting to an Abnormal TCD Velocity in Children With Sickle Cell Anemia and Conditional Pre-treatment TCD Velocities.
Brief Title: Sparing Conversion to Abnormal TCD (Transcranial Doppler) Elevation (SCATE)
Acronym: SCATE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: inability to reach a satisfactory endpoint with respect to adequate recruitment
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); St. Jude Children's Research Hospital (Other); Tropical Medicine Research Institute (Other); Instituto Estadual de Hematologia Arthur de Siqueira Cavalcanti (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-29205 SCATE; R01HL098239 (NIH)
Record Dates: First submitted 2012-02-06; First posted 2012-02-13 (Estimated); Results first posted 2015-12-09 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Sickle Cell Anemia
Keywords: Phase III; Sickle cell anemia; Conditional transcranial doppler velocities; Reduce risk of conversion to abnormally high transcranial doppler velocities; Pediatric patients
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Therapy: Observation (No Intervention): Half of the subjects will be randomized to clinical observation only, which includes monthly visits with clinical evaluations, laboratory tests, and TCD endpoint examinations
- Hydroxyurea (Experimental): Half of the subjects will be randomized to hydroxyurea, taken as capsules (300 mg, 400 mg, or 500 mg), or as a liquid formulation (100 mg/mL). Hydroxyurea will be administered once daily by mouth. Subjects will be monitored monthly with clinical evaluations, laboratory tests, and TCD endpoint examinations.
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea — Hydroxyurea will be administered once daily, in either capsule form (300mg, 400mg, or 500mg) or as a liquid formulation (100mg/ml). Dosing will commence at 20 mg/kg/day. Dose escalation will occur in 5 mg/kg/day increments, adjusting every 8 weeks unless hematological toxicity occurs.
  Other Names: Hydroxycarbamide; Hydrea; Droxia
  Arms: Hydroxyurea

SUMMARY:
The primary goal of the Phase III SCATE trial is to compare 30 months of alternative therapy (hydroxyurea) to standard care (observation) in children with sickle cell anemia and conditional (170 - 199cm/sec) Transcranial Doppler (TCD) velocities. For the alternative regimen (hydroxyurea) to be declared superior to the standard treatment regimen (observation), the hydroxyurea-treated group must have a three-fold reduction in the incidence of conversion to abnormal TCD velocities (≥ 200 cm/sec), compared to the standard treatment arm.

DETAILED DESCRIPTION:
Results from previous studies confirm an increased risk of stroke among children with conditional TCD velocities. In addition, studies suggest that patients who were on observation alone, converted from conditional TCD (moderate risk category) to an abnormal TCD (with a much higher risk for primary stroke) within 30 months of initial identification of the conditional TCD velocity; this conversion led to initiation of chronic and indefinite transfusions in all cases. Preliminary data suggests that the risk of conversion to abnormal TCD velocities will be lower for subjects with conditional TCD velocities on hydroxyurea by at least three-fold. This important difference in conversion risk rate suggests that an alternative treatment could have a substantial and beneficial impact on patients with elevated TCD velocities.

An alternative treatment could protect the brain of patients with SCA and conditional TCD velocities who are at increased risk for stroke. The avoidance of chronic blood transfusions would be a great benefit for all children with sickle cell disease, especially those in developing countries where the blood supply may be less safe (in comparison with that in the US) or unavailable, and very costly.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric subjects with severe forms of sickle cell anemia (HbSS, HbSβ0 thalassemia, HbSD, HbSOArab)
2. Age: ≥ 2 and < 11 years of age, at the time of enrollment
3. Conditional TCD Velocity (170 - 199cm/sec) by Transcranial Doppler ultrasonography examination within 3 months of enrollment
4. Parent or guardian willing and able to provide informed consent
5. Ability to comply with study related treatments, evaluations, and follow-up

Exclusion Criteria:

1. Prior abnormal TCD Velocity
2. History of clinical stroke
3. Inability to take or tolerate daily oral hydroxyurea, including

   * Known allergy to hydroxyurea therapy
   * Known positive serology to HIV infection
   * Known malignancy
   * Current lactation
4. Abnormal laboratory values at initial evaluation (temporary exclusions):

   * Hemoglobin concentration < 6.0 gm/dL
   * Absolute reticulocyte count < 100 x 10^9/L with a hemoglobin concentration < 8.0 gm/dL
   * WBC count < 3.0 x 10^9/L
   * Absolute neutrophil count (ANC) < 1.0 x 10^9/L
   * Platelet count < 100 x 10^9/L
5. Current use of therapeutic agents for sickle cell disease (e.g., hydroxyurea, arginine, decitabine, magnesium, chronic transfusions). Subjects must be off therapeutic agents for sickle cell disease for at least 3 months prior to enrollment.
6. Current participation in other therapeutic clinical trials
7. Serum creatinine more than twice the upper limit for age OR ≥ 1.0 mg/dL
8. Any condition or chronic illness, which in the opinion of the clinical investigator makes participation ill-advised
9. Pregnancy (for post-menarchal females only)
10. Erythrocyte transfusion within the past 2 months
11. Previous stem cell transplant or other myelosuppressive therapy

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2012-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell E. Ware, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (3):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States
- Instituto Estadual de Hematologia Arthur de Siqueira Cavalcanti (HEMORIO), Centro, Rio de Janeiro, Brazil
- Tropical Medicine Research Institute, University of the West Indies (UWI), Mona, Kingston, Jamaica

REFERENCES:
- [Result] Hankins JS, McCarville MB, Rankine-Mullings A, Reid ME, Lobo CL, Moura PG, Ali S, Soares DP, Aldred K, Jay DW, Aygun B, Bennett J, Kang G, Goldsmith JC, Smeltzer MP, Boyett JM, Ware RE. Prevention of conversion to abnormal transcranial Doppler with hydroxyurea in sickle cell anemia: A Phase III international randomized clinical trial. Am J Hematol. 2015 Dec;90(12):1099-105. doi: 10.1002/ajh.24198. Epub 2015 Nov 17. PMID 26414435

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 22 participants were randomized (e.g., a total of 38 participants enrolled, but only 22 participants were randomized to treatment)
Period: Overall Study
Arm/Group | Hydroxyurea | Standard Therapy: Observation
Started | 11 | 11
Completed | 0 | 0
Not Completed | 11 | 11
Not completed — Early termination of study | 11 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Therapy: Observation | Hydroxyurea | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 11 | 22
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 6.3 (1.5) | 6 (2.4) | 6.15 (1.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  Jamaica | 7 | 6 | 13
  Brazil | 2 | 3 | 5
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Conversion to Abnormal Maximum TAMV
Description: The primary endpoint of the SCATE trial is the cumulative incidence of conversion to abnormal maximum TAMV (time-averaged mean velocity) measured by transcranial doppler (TCD) ultrasonography. Subjects must have conditional velocities at baseline, defined as 170 - 199 cm/sec, which indicate moderate stroke risk. Abnormal velocities are defined as ≥ 200 cm/sec, which indicate high stroke risk. The number of conversions from conditional velocities to abnormal velocities in each treatment arm will be compared as the primary outcome.
Time Frame: 30 months
Population: No participants reached 30 months of treatment prior to study termination; therefore, the primary outcome measure was not analyzed.
Arm/Group | Hydroxyurea | Standard Therapy: Observation
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Serial TCD Velocities
Description: This secondary outcome measure will be the highest TAMV obtained in specific arteries. Serial TCD velocities are measured throughout the SCATE trial and will be compared to the baseline value.
Time Frame: 30 months
Population: No participants reached 30 months of treatment prior to study termination; therefore, the secondary outcome measures were not analyzed.
Arm/Group | Hydroxyurea | Standard Therapy: Observation
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Cumulative Incidence of Neurological Events
Description: The cumulative incidence of neurological events as a secondary endpoint, which include both stroke and non-stroke neurological events, will be determined over the treatment period for both standard and alternative arms.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Hydroxyurea | Standard Therapy: Observation
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Cumulative Incidence of Non-Neurological Events
Description: The cumulative incidence of non-neurological sickle cell-related events, including vaso-occlusion and splenic sequestration, will be estimated over the treatment period for both standard and alternative arms.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Hydroxyurea | Standard Therapy: Observation
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Quality of Life
Description: Standard Quality of Life measure will be taken during specific time points, as well as one newly-developed Sickle Cell Disease Quality of Life measure.
Time Frame: 30 months
Population: as for outcome 2
Arm/Group | Hydroxyurea | Standard Therapy: Observation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: May 2012 - Jan 2014 = 20 months
Description: AEs below grade 2 were not recorded for the SCATE trial
Arm/Group | Hydroxyurea | Standard Therapy: Observation
Serious Adverse Events (participants affected / at risk) | 6/11 | 11/11
Other Adverse Events (participants affected / at risk) | 7/11 | 7/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxyurea (N=11) | Standard Therapy: Observation (N=11)
Hemoglobin (Blood and lymphatic system disorders) | 1 (11) | 3 (11)
Fever (General disorders) | 1 (11) | 0 (0)
Hepatobiliary Disorder (Hepatobiliary disorders) | 2 (11) | 0 (0)
Infections and Infestations (Infections and infestations) | 1 (11) | 0 (0)
Lung Infection (Infections and infestations) | 0 (0) | 1 (11)
Lymph gland infection (Infections and infestations) | 0 (0) | 1 (11)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (11)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (11)
Acute Chest Syndrome (General disorders) | 0 (0) | 1 (11)
Acute Splenic Sequestration (General disorders) | 1 (11) | 1 (11)
Vaso-occlusive Event (General disorders) | 0 (0) | 1 (11)
AST (General disorders) | 1 (11) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (11)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxyurea (N=11) | Standard Therapy: Observation (N=11)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 2 (2) | 2 (2)
Flu Like Symptoms (General disorders) | 1 (1) | 1 (1)
Non Cardiac Chest Pain (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Hepatobiliary Disorders (Hepatobiliary disorders) | 1 (1) | 0 (0)
Infections and Infestations (Infections and infestations) | 1 (1) | 1 (1)
Lung infections (Infections and infestations) | 0 (0) | 1 (1)
Lymph Glad Infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth Infection (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 2 (2) | 1 (1)
Metabolism and Nutrition Disorders (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 2 (2)
Dysnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute Chest Syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute Stlenic sequestration (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Vaso-occlusive Event (Blood and lymphatic system disorders) | 2 (2) | 3 (4)
ANC (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ARC (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
AST (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 2 (3)
Bilirubin (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Skin and subcutaneous tissue dissorder other (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No